CLINICAL TRIAL: NCT04396548
Title: Preoperative Midodrine for Improving Hemodynamics in Orthopedic Patients Undergoing Spinal Anesthesia
Brief Title: Midodrine for Improving Hemodynamics After Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohammed Alseoudy, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Midodrine and SA
Record Dates: First submitted 2020-05-16; First posted 2020-05-20 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Hypotension After Spinal Anesthesia
Keywords: midodrine before spinal anesthesia
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: The study subjects and the resident assessing the outcomes will be blinded to the study group. A single investigator will assess the patients for eligibility, obtain written informed consent, open the sealed opaque envelopes containing group allocation and administer oral tablet.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (midodrine group) (Active Comparator): Midodrine will be given orally with small sips of water one hour before arrival in the operation room before spinal anesthesia
  Interventions: Drug: Midodrine Oral Product
- Group B (placebo group): (Placebo Comparator): Inert tablet containing sugar (placebo) will be given orally with small sips of water one hour before arrival in the operation room before spinal anesthesia
  Interventions: Drug: Inert tablet containing sugar (placebo)

INTERVENTIONS:
Drug: Midodrine Oral Product — Patients will receive oral 10 mg tablet of midodrine with small sips of water one hour before arrival in the operation room. All patients will be monitored in with noninvasive blood pressure as well as continuous electrocardiogram (ECG) and pulse oximetry (SpO2). Before placement of spinal anesthesia, all patients will receive an IV bolus of 10mL/kg of Lactated Ringer's . Spinal anesthesia (midline puncture) will be performed in sitting position by a staff anesthetist at L3-L4 or L4-L5 with a 25-gauge Withacre needle injecting 12.5 mg of hyperbaric 0.5% bupivacaine (2.5 mL) with 10μg fentanyl. After injection,the patients will be turned supine.
  Other Names: spinal anesthesia
  Arms: Group A (midodrine group)
Drug: Inert tablet containing sugar (placebo) — : Patients will receive Inert tablet containing sugar (placebo) with small sips of water one hour before arrival in the operation room. All patients will be monitored in with noninvasive blood pressure as well as continuous electrocardiogram (ECG) and pulse oximetry (SpO2). Before placement of spinal anesthesia, all patients will receive an IV bolus of 10mL/kg of Lactated Ringer's . Spinal anesthesia (midline puncture) will be performed in sitting position by a staff anesthetist at L3-L4 or L4-L5 with a 25-gauge Withacre needle injecting 12.5 mg of hyperbaric 0.5% bupivacaine (2.5 mL) with 10μg fentanyl. After injection,the patients will be turned supine
  Other Names: spinal anesthesia
  Arms: Group B (placebo group):

SUMMARY:
Neuraxial blockade such as spinal anaesthesia can cause severe hypotension due to pharmacological sympathectomy resulting in potential deleterious consequences for the patient. Prevention of this spinal anaesthesia induced hypotension is of utmost importance. Techniques currently in use for preventing hypotension include intravenous fluid prehydration, sympathomimetic drugs, and physical methods such as leg bindings and compression stockings. Midodrine is a direct acting α1-adrenoceptor agonist which causes venous and arterial vasoconstriction through stimulation of α1- receptors located in the vasculature. The aim of this study is to evaluate the efficacy and safety of prophylactic midodrine use with preoperative fluid hydration before spinal anesthesia in the prevention of hypotension in patients undergoing elective orthopedic surgery. We hypothesize that intraoperative hypotension would be less in patients given midodrine and intravenous fluid prehydration preoperatively before spinal anesthesia.

DETAILED DESCRIPTION:
Neuraxial blockade such as spinal anaesthesia can cause severe hypotension due to pharmacological sympathectomy resulting in potential deleterious consequences for the patient. Prevention of this spinal anaesthesia induced hypotension is of utmost importance. Several techniques and methodologies have been adopted for the prevention of this neuraxial hypotension with varying degree of success. Techniques currently in use for preventing hypotension include intravenous fluid prehydration, sympathomimetic drugs, and physical methods such as leg bindings and compression stockings. Midodrine is a direct acting α1-adrenoceptor agonist which causes venous and arterial vasoconstriction through stimulation of α1- receptors located in the vasculature. The net result is an increase in vascular tone and systolic blood pressure. Cardiac β-receptors are unaffected and there is no significant blood brain barrier penetration. We hypothesize that intraoperative hypotension would be less in patients given midodrine and intravenous fluid prehydration preoperatively before spinal anesthesia. The study will include 80 patients who will be scheduled for elective orthopedic surgery on the lower extremities undergoing spinal anesthesia. It will be conducted in Mansoura University Hospital after getting approval from Institutional Review Board (IRB), Faculty of medicine, Mansoura University. Informed written consents will be obtained from all subjects in the study after ensuring confidentiality. Patients will be randomly allocated using computer generated random numbers to either treatment with midodrine (group M) or control (group C) using the sealed opaque envelope technique. Patients in group M will receive oral 10 mg tablet of midodrine with small sips of water one hour before arrival in the operation room while patients in group C will receive inert tablet containing sugar (placebo) at the same time. All patients will be monitored in with noninvasive blood pressure as well ascontinuous electrocardiogram (ECG) and pulse oximetry (SpO2). Before placement of spinal anesthesia, all patients will receive an IV bolus of 10mL/kg of Lactated Ringer's. Spinal anesthesia (midline puncture) will be performed in sitting position by a staff anesthetist at L3-L4 or L4-L5 with a 25-gauge Withacre needle injecting 12.5 mg of hyperbaric 0.5% bupivacaine (2.5 mL) with 10μg fentanyl. After injection,the patients will be turned supine. The baseline arterial blood pressure (mean) will be calculated as the average of 3 consecutive measurements before placement of the SA every 15 min after taking midodrine and every 5 min for 30 min after spinal anesthesia. Any vasovagal syncopes will be recorded. After placement of the SA, the patient's heart rate will be obtained every five minutes for 30 minutes and thereafter, in accordance with standard clinical practice, every 5 minutes until the end of surgery. The dermatome level of the sensory block using loss of pinprick will be checked every 5 minutes for 20minutes. The modified Bromage scale (0 = no motor block, 1 = straight leg hip flexion blocked, 2 = knee flexion blocked, 3 = complete motor block) will be used to quantify the degree of motor block at 20 minutes. Reqirements of ephedrine and atropine and fluide intake will be recorded. time to onset of the first hypotension, the proportion of patients without hypotension, and the number of bradycardic episodes per patient will also be recorded. Perioperative copmlications such as reactive hypertension, nausea, vomiting, hypothermia, shivering and postdural puncture headache will be recorded. An investigator who is blind to type of intervention wil be responsible for collection of data.

ELIGIBILITY:
Inclusion Criteria:

* • American Society of Anesthesiologists (ASA) status: 1 or 2 .

  * Orthopedic surgery on the lower extremities

Exclusion Criteria:

* • Pheochromocytoma. .Throtoxicosis. .Structural heart disease.

  * Baseline blood pressure more than 140/90 .Acute kidney failure.
  * Any contraindications to spinal anesthesia such as local infection and coagulopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
1. incidence perioperative hypotension | Up to 4 hours after surgery
  the number of hypotensive patients will be recorded

SECONDARY OUTCOMES:
change in mean arterial blood pressure | Up to 4 hours after surgery
  Mean arterial blood pressure will be recorded basal and every 15 min after taking midodrine and every 5 min after spinal anesthesia till end of surgery and every
change in heart rate | Up to 4 hours after surgery
  heart rate will be recorded basal and every 15 min after taking midodrine and every 5 min after spinal anesthesia till end of surgery and every 15 minutes after surgery
requirements of ephedrine and atropine | Up to 4 hours after the procedure
  amount of ephedrine and atropine to treat hypotension and bradycardia
incidence of adverse effects | Up to 24 hours surgery
  nausea, vomiting, shivering and postdural puncture headache will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M Alseoudy, MD, Principal Investigator — Faculty of Medicine, Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alseoudy MM, Nasr MO, Abdelsalam TA. Efficacy of Preoperative Oral Midodrine in Preventing Hypotension After Spinal Anesthesia in Young Adults: A Randomized Controlled Trial. Anesth Analg. 2022 Nov 1;135(5):1089-1096. doi: 10.1213/ANE.0000000000006173. Epub 2022 Aug 10. PMID 35950781